CLINICAL TRIAL: NCT04027790
Title: Clinical Sample Protocol for Plasma-based Colorectal Cancer Screening Research & Development
Brief Title: Plasma-based Colorectal Cancer Screening Research & Development
Status: Completed | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ECS0001
Record Dates: First submitted 2019-06-06; First posted 2019-07-22 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Colo-rectal Cancer
Keywords: plasma; cell-free DNA; DNA Methylation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1 - Cancer Patients: Subjects with known colorectal cancer (i.e. AJCC/UICC stages 0, I, II, and III) who provide plasma at least 7 days after diagnosis by colonoscopy, but prior to surgery or treatment
  Interventions: Diagnostic Test: Epi proColon
- Group 2 - Screening Subjects: Prospectively enrolled subjects reporting for screening colonoscopy who provide a blood sample up to 2 weeks prior to bowel prep and prior to colonoscopy. We accept all subjects who meet the institutional criteria as average risk subjects referred for a screening colonoscopy for colorectal cancer, including subjects undergoing a colonoscopy as a follow-up to a positive (non-colonoscopic) test
  Interventions: Diagnostic Test: Epi proColon

INTERVENTIONS:
Diagnostic Test: Epi proColon — Analysis of DNA methylation status for Septin9 and additional biomarkers

SUMMARY:
The objective of this Clinical Sample Collection Study is to develop a biobank of appropriately collected plasma samples from colorectal cancer patients (i.e. AJCC/UICC stages 0, I, II, III) prior to therapeutic intervention, and from people reporting for colorectal cancer screening by colonoscopy, prior to bowel preparation.

DETAILED DESCRIPTION:
The objective of this Clinical Sample Collection Study is to develop a biobank of appropriately collected plasma samples from colorectal cancer patients (i.e. AJCC/UICC stages 0, I, II, III) prior to therapeutic intervention, and from people reporting for colorectal cancer screening by colonoscopy, prior to bowel preparation. Samples in the colorectal cancer biobank will be used to: 1) assess the clinical performance of novel biomarkers for colorectal cancer screening; 2) develop improved processing workflows for the Epi proColon® test; 3) develop an automated Epi BiSKit workflow.

ELIGIBILITY:
Inclusion Criteria: Group 1

* Willing and able to sign an Informed Consent and adhere to study requirements.
* Subjects with colorectal cancer preferably detected by screening (any guideline recommended modality).
* Colonoscopy diagnosis of colorectal cancer (CRC).*
* Blood sampling a minimum of 7 days after colonoscopy and before resection surgery.

  * = Strong clinical suspicion of colorectal carcinoma is also acceptable for subject enrollment; Case must have a confirmed diagnosis after surgery of CRC and be accompanied by a complete final pathology report.

Inclusion Criteria: Group 2

* Willing and able to sign an Informed Consent and adhere to study requirements.
* Eligible for colorectal cancer screening colonoscopy.
* 45 - 84 years of age at blood sampling.
* Able to provide blood sample within up to 2 weeks prior to bowel prep and colonoscopy.

Exclusion Criteria: Group 1

* Subject with curative biopsy during colonoscopy.
* Current neoadjuvant treatment.
* Current diagnosis of any cancer other than CRC, except non-melanoma skin cancer.
* Known infection with HIV, HBV or HCV.

Exclusion Criteria: Group 2

* Previous personal history of CRC, adenomatous polyps >10mm or sessile serrated adenomas (polyps).
* Familial risk for colorectal cancer (1 or more 1st degree relatives with CRC; known HNPCC or FAP).
* History of inflammatory bowel disease.
* Current neoadjuvant treatment.
* Current diagnosis of any cancer other than CRC, except non-melanoma skin cancer.
* infection with HIV, HBV or HCV.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women and Men age 45-84 reporting for screening colonoscopy (Group 2) or with known colorectal cancer, prior to intervention (Group 1).
Sampling Method: Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Test Positivity | Anticipated time frame for testing blood sample is within 12 months of collection
  DNA methylation status of Epi proColon and biomarker panel

CONTACTS AND LOCATIONS:
Overall Officials: Theo deVos, PhD, Study Director — Epigenomics, Inc
Locations (5):
- United States (5):
  - University of South Florida, Tampa, Florida
  - Springfield Clinic, Springfield, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington University, St Louis, Missouri
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania